CLINICAL TRIAL: NCT01745458
Title: A Double Blind Study to Evaluate Effects of Repeat Doses of SB-659032 on Platelet Aggregation in Healthy Volunteers
Brief Title: SB-659032 Platelet Aggregation Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 104623
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — rilapladib

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- SB-659032 (Experimental): 250 mg non-enteric coated SB-659032
  Interventions: Drug: Placebo
- Placebo (Placebo Comparator): matched placebo QD for 14 days
  Interventions: Drug: SB-659032

INTERVENTIONS:
Drug: SB-659032
  Arms: Placebo
Drug: Placebo — Matched placebo
  Arms: SB-659032

SUMMARY:
This study is designed to assess whether inhibition of plasma Lp-PLA2 activity impacts platelet function as assessed by ex vivo platelet aggregation tests and in vivo plasma biomarkers.

DETAILED DESCRIPTION:
SB-659032 is a selective and orally active inhibitor of lipoprotein-associated phospholipase A2 (Lp-PLA2) that is being developed for the treatment of atherosclerosis. This study is designed to assess whether inhibition of plasma Lp-PLA2 activity impacts platelet function as assessed by ex vivo platelet aggregation tests and in vivo plasma biomarkers. Blood samples for PK analysis and measurement of Lp-PLA2 activity will also be collected. Questionnaires will be completed to evaluate the frequency of odorrelated AEs with non-enteric coated formulation of SB-659032 relative to placebo. This will be a double blind, repeat dose, randomized, placebo-controlled, two period, period balanced, crossover study. There will be a minimum of a 21 day washout period between dosing in each period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males between 18 and 55 years of age, inclusive
* Body weight greater than 50 kg (110 pounds) and body mass index (BMI) between 19 and 32 where: BMI = weight in kg/(height in meters)2
* A signed and dated written informed consent prior to admission to the study
* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Any clinically relevant abnormality identified on the screening medical assessment, laboratory examination or ECG
* Platelet count below or above the reference range
* History of hypercoagulable state or history of thrombosis
* History of platelet dysfunction
* A known history of Gilbert's Syndrome
* History of asthma, anaphylaxis or anaphalactoid reactions, severe allergic responses
* A history of alcohol, substance or drug abuse within the last year or a positive alcohol breath test at screening or predose in each period. Abuse of alcohol is defined as an average weekly intake of greater than or equal to 21 units (male) or an average daily intake of greater than or equal to 3 units (male). 1 unit is equivalent to a 285mL glass of full strength beer or 425 mL schooner of light beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine
* Positive urine drug screen at screening or predose in each period
* History of use of tobacco or nicotine containing products within 6 months of screening or a positive urine cotinine at screening or exhaled carbon monoxide test at predose in each period
* Positive HIV, Hepatitis B or Hepatitis C at screening
* Use of aspirin, aspirin-containing products, non-steroidal anti-inflammatory agents or any antiplatelet medication within 14 days prior to Day -1 of the study (a list of these drugs will be reviewed with the subject at screening and provided to them to take home)
* Use of prescription (including hormone replacement therapy) or non-prescription drugs and vitamins within 7 days or 5 half-lives (whichever is longer) prior to Day -1 of the study. An exception is acetaminophen which is allowed at doses of ≤ 2g/day
* Use of dietary/herbal supplements including (but not limited to) St. John's wort, kava, ephedra (ma huang), gingko biloba, DHEA, yohimbe, saw palmetto, ginseng and red yeast rice within 14 days prior to Day -1 of the study
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to dosing
* Consumption of grapefruit or grapefruit juice within 7 days prior to Day -1 of the study
* A history of cholecystectomy or biliary tract disease including a history of liver disease with elevated liver function tests of known or unknown etiology
* An unwillingness to abstain from sexual intercourse with pregnant or lactating women or an unwillingness to use a condom and another form of contraception (e.g., IUD, birth control pills taken by female partner, diaphragm with spermicide) if engaging in sexual intercourse with a woman who could become pregnant until discharge from the study
* Donation of blood in excess of 500 mL within 56 days or donation of blood in excess of 250 mL within 7 days prior to dosing
* Full ADP- and/or collagen-induced aggregation (greater than and equal to 40%) at all three concentrations of one or both agonists, as assessed within 6 months prior to first dose and at Day -1 of each period
* No ADP- or collagen-induced aggregation (less than 40%) at the highest concentration of either agonist, as assessed within 6 months prior to first dose and at Day -1 of each period

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2005-07; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation | 14 days
  Percent maximum platelet aggregation following ADP- and collagen-induced aggregation
Biomarkers of platelet aggregation | 14 days
  Urinary 11-dehydrothromboxane B2 and blood CD62 concentrations

SECONDARY OUTCOMES:
Lp-PLA2 inhibition | 14 days
  Lp-PLA2 activity, expressed in terms of percent inhibition relative to baseline
Clinical safety data | 14 days
  spontaneous adverse event reporting, 12-Lead ECG, vital signs, nursing/physician observation and safety and laboratory tests
Mean concentrations of SB-659032 and its major metabolite, SB-664601 | 14 days
  SB-659032 and SB-664601 concentrations
Frequency and intensity of odor-related adverse events | 14 days
  The frequency and intensity of odor-related adverse events as reported by subjects will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Shaddinger BC, Xu Y, Roger JH, Macphee CH, Handel M, Baidoo CA, Magee M, Lepore JJ, Sprecher DL. Platelet aggregation unchanged by lipoprotein-associated phospholipase A(2) inhibition: results from an in vitro study and two randomized phase I trials. PLoS One. 2014 Jan 27;9(1):e83094. doi: 10.1371/journal.pone.0083094. eCollection 2014. PMID 24475026